CLINICAL TRIAL: NCT01887249
Title: Randomized Clinical Trial: the Comparison of 15-day Sequential and 10-day Sequential Therapy to PPI-based Triple Therapy for Helicobacter Pylori Infection in Korea
Brief Title: 15-day Sequential Therapy for Helicobacter Pylori Infection in Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ministry of Education, Republic of Korea (2012R1A1A3A04002680) (Unknown)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, M.D., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1007/106-001
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Clarithromycin; Metronidazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 15 day sequential eradication therapy (Experimental): the 15-day sequential therapy regimen, which consisted of esomeprazole (40 mg) plus amoxicillin (1000 mg) twice a day for 5 days, then esomeprazole (40 mg) with clarithromycin (500 mg) and metronidazole (500 mg) twice a day for 10 days.
  Interventions: Drug: Clarithromycin; Drug: metronidazole; Drug: esomeprazole
- 10-day sequential eradication therapy (Active Comparator): the 10-day sequential therapy regimen, which consisted of esomeprazole (40 mg) plus amoxicillin (1000 mg) twice a day for 5 days, then esomeprazole (40 mg) with clarithromycin (500 mg) and metronidazole (500 mg) twice a day for another five days
  Interventions: Drug: Clarithromycin; Drug: metronidazole; Drug: esomeprazole
- 7-day PPI triple eradication therapy (No Intervention): 7-day PPI triple therapy regimen, which consisted of esomeprazole (40mg) plus amoxicillin (1000mg) and clarithromycin (500mg) twice daily for 7 days.

INTERVENTIONS:
Drug: Clarithromycin
  Arms: 10-day sequential eradication therapy; 15 day sequential eradication therapy
Drug: metronidazole
  Arms: 10-day sequential eradication therapy; 15 day sequential eradication therapy
Drug: esomeprazole
  Arms: 10-day sequential eradication therapy; 15 day sequential eradication therapy

SUMMARY:
10-day sequential therapy was not sufficient to overcome tough situation for H. pylori eradication in Korea due to high antimicrobial resistance. The present investigators assumed that doubling duration of second phase of sequential therapy might have more potent bactericidal efficacy than previous 10-day sequential regimen. But 15-day regimen with initial 5-day PPI with amoxicillin followed by remaining 10-day PPI, clarithromycin with metronidazole was not ever tested before. Moreover, whether extending the sequential therapy to 15-day might be more effective than 10-day sequential therapy is unknown especially in Korea. From this background, the present investigators prepared clinical trials regarding modified sequential therapy which was extending the treatment duration to 15 days compared than previous 10-day sequential therapy regimen. In addition, pre-treatment antimicrobial susceptibility testing was performed to find the possibility to overcome antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* patients with H. pylori infection who had never received treatment for H. pylori infection
* H. pylori infection defined by a positive rapid urease test (CLOtest, Delta West, Bentley, Australia) by gastric mucosal biopsy from the lesser curvature of the mid antrum or mid body or histological evidence of H. pylori by modified Giemsa staining in the lesser and greater curvature of the mid antrum or mid body, respectively or a positive C-urea breath test.

Exclusion Criteria:

* Patients with concurrent critical illness, a history of previous upper gastrointestinal surgery, contraindication to any of the study medications, recent frequent intake of NSAIDs, anticoagulants or steroids, an allergy to the study medications, and those that were pregnant or breast-feeding women were excluded from the study. Other exclusion criteria include recent use of antimicrobials and any condition probably associated with poor compliance such as drug abusers or alcoholics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2010-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Four weeks after completing eradication therapy

SECONDARY OUTCOMES:
Frequency and severity of side effects, Drug Compliance | Four weeks after completing eradication therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Bundang-gu, Seongnam, Gyeonggi-do, South Korea